CLINICAL TRIAL: NCT04522752
Title: Long-term Endoscopic Follow-up of Benign Epithelial Gastric Polyps: a Multicenter Prospective Large Sample Cohort Study
Brief Title: Long-term Endoscopic Follow-up of Benign Epithelial Gastric Polyps
Acronym: LEFBEGP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Other Study IDs: XJTU1AF-CRF-2018-016
Record Dates: First submitted 2020-08-19; First posted 2020-08-21 (Actual); Last update posted 2022-05-09 (Actual); Status verified 2021-08

CONDITIONS: Benign Gastric Polyp
Keywords: benign gastric polyp; gastroendoscopy; pathological type

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsy of benign epithelial gastric polyps
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Gastric Polyp: The included subjects were patients with benign epithelial gastric polyps confirmed by gastroscopy and biopsy pathology. The size and pathology type of polyps were identified. Gastroscopy and biopsy were followed up six, twelve and eighteen months later to observe the relationship between the size, pathology types of polyps and the development of gastric polyps. Other factors including the relationship between helicobacter pylori infection and polyp type were also observed.
  Interventions: Other: Size and pathological type of benign epithelial gastric polyp

INTERVENTIONS:
Other: Size and pathological type of benign epithelial gastric polyp — All subjects will undergo gastroscopy and biopsy to determine the size and pathological type of benign epithelial gastric polyps.The correlation between polyp size and type and polyp development was observed at 6 months, 12 months and 18 months after inclusion.

SUMMARY:
Benign epithelial gastric polyps are benign raised lesions that originate from the gastric mucosa or submucosa and protrude from the gastric cavity with a wide base or a pedicle.The diagnosis and treatment of benign epithelial gastric polyps are currently controversial. There is still a lack of clinical research evidence especially for the malignant tendency and related treatments of gastric polyps. Many doctors have ambiguous understanding of benign epithelial gastric polyps and their endoscopic management is still in a"one size fits all"mode in China, which greatly wastes medical resources and increases the medical risks of patients, So it is imminent to formulate management practices for the diagnosis and treatment of gastric polyps. Therefore, a full understanding of the clinical characteristics, endoscopic characteristics and long-term follow-up trends of benign epithelial gastric polyps is of great significance for clinicians to formulate reasonable treatment and follow-up plans. This study is a prospective, large-sample observational cohort study. It is planned to include 200 patients with biopsy confirmed benign epithelial gastric polyps participating in this study from September 10, 2020 to December 31, 2021 and followed up for 18 months. The main research endpoint is the correlation between size and pathological type of benign epithelial gastric polyps and polyps development. The secondary research endpoint is the correlation between type of benign epithelial gastric polyps and Helicobacter pylori infection. The research results will help provide long-term follow-up data for benign epithelial gastric polyps of different pathological types, thereby providing first-hand evidence-based medical data for formulating gastric polyp management guidelines, helping to efficiently screen high-risk groups and guiding their examination, treatment and long-term follow-up to achieve early detection and early treatment of gastric cancer, thereby reducing the mortality rate.

ELIGIBILITY:
Inclusion Criteria:

* After gastroscopy, gastric polyps are found and pathological biopsy is obtained.

All polyps undergo endoscopic clamp biopsy, requiring at least one piece of tissue from each polyp to be submitted for examination.

Exclusion Criteria:

* Submucosal raised lesions.
* Gastrointestinal bleeding.
* Concomitant with gastric malignant tumor disease or previous gastric surgery for any reason.
* Benign polyps with a diameter greater than 1cm, regardless of the pathological type.
* The patient also has other serious diseases that affect the evaluation of this study, such as severe liver disease, heart disease, kidney disease, malignant tumors and alcoholism.
* The patient cannot express his main complaint correctly, such as mental illness, severe neurosis, and cannot cooperate with the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The subjects of this study are 18 to 70 years old patients who underwent gastroscopy from September 10, 2020 to December 31, 2021 and were confirmed by biopsy to be benign epithelial gastric polyps patients. At the same time, there are no exclusion criteria for the research objects.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-30 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2023-09-10 (Estimated)

PRIMARY OUTCOMES:
Correlation between size and pathological type of benign epithelial gastric polyp and polyp development. | The planned observation period of this study is 18 months.
  Gastroscopy and pathological examination were performed at 6, 12, and 18 months after inclusion to observe the correlation between size and pathological type of benign epithelial gastric polyps and polyp development.

SECONDARY OUTCOMES:
Correlation between helicobacter pylori infection and pathological type of benign epithelial gastric polyp. | The planned observation period of this study is 18 months.
  To investigate the infection status of the subjects with Helicobacter pylori and analyze its correlation with the pathological types of benign epithelial gastric polyps.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxia Li, M.D., Principal Investigator — First Affiliated Hospital Xi'an Jiaotong University
Locations (1):
- First Affliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: Yes
We plan to share individual participant data with relevant industry researchers.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: The data will be open and shared by December 2022 for three years.
Access Criteria: Registered and certified medical researchers.

REFERENCES:
- [Result] Schmitz JM, Stolte M. Gastric polyps as precancerous lesions. Gastrointest Endosc Clin N Am. 1997 Jan;7(1):29-46. PMID 8995111
- [Result] Dinis-Ribeiro M, Areia M, de Vries AC, Marcos-Pinto R, Monteiro-Soares M, O'Connor A, Pereira C, Pimentel-Nunes P, Correia R, Ensari A, Dumonceau JM, Machado JC, Macedo G, Malfertheiner P, Matysiak-Budnik T, Megraud F, Miki K, O'Morain C, Peek RM, Ponchon T, Ristimaki A, Rembacken B, Carneiro F, Kuipers EJ; European Society of Gastrointestinal Endoscopy; European Helicobacter Study Group; European Society of Pathology; Sociedade Portuguesa de Endoscopia Digestiva. Management of precancerous conditions and lesions in the stomach (MAPS): guideline from the European Society of Gastrointestinal Endoscopy (ESGE), European Helicobacter Study Group (EHSG), European Society of Pathology (ESP), and the Sociedade Portuguesa de Endoscopia Digestiva (SPED). Endoscopy. 2012 Jan;44(1):74-94. doi: 10.1055/s-0031-1291491. Epub 2011 Dec 23. PMID 22198778
- [Result] Jalving M, Koornstra JJ, Wesseling J, Boezen HM, DE Jong S, Kleibeuker JH. Increased risk of fundic gland polyps during long-term proton pump inhibitor therapy. Aliment Pharmacol Ther. 2006 Nov 1;24(9):1341-8. doi: 10.1111/j.1365-2036.2006.03127.x. PMID 17059515
- [Result] Genta RM, Schuler CM, Robiou CI, Lash RH. No association between gastric fundic gland polyps and gastrointestinal neoplasia in a study of over 100,000 patients. Clin Gastroenterol Hepatol. 2009 Aug;7(8):849-54. doi: 10.1016/j.cgh.2009.05.015. Epub 2009 May 22. PMID 19465154
- [Result] Tran-Duy A, Spaetgens B, Hoes AW, de Wit NJ, Stehouwer CD. Use of Proton Pump Inhibitors and Risks of Fundic Gland Polyps and Gastric Cancer: Systematic Review and Meta-analysis. Clin Gastroenterol Hepatol. 2016 Dec;14(12):1706-1719.e5. doi: 10.1016/j.cgh.2016.05.018. Epub 2016 May 20. PMID 27211501
- [Result] Hirota WK, Zuckerman MJ, Adler DG, Davila RE, Egan J, Leighton JA, Qureshi WA, Rajan E, Fanelli R, Wheeler-Harbaugh J, Baron TH, Faigel DO; Standards of Practice Committee, American Society for Gastrointestinal Endoscopy. ASGE guideline: the role of endoscopy in the surveillance of premalignant conditions of the upper GI tract. Gastrointest Endosc. 2006 Apr;63(4):570-80. doi: 10.1016/j.gie.2006.02.004. No abstract available. PMID 16564854